CLINICAL TRIAL: NCT03294512
Title: Pilot and Feasibility Study of a MAWDS (Medications, Activity, Weight, Diet and Symptoms) Heart Failure Mobile Platform (iMAWDS Mobile HF Study)
Brief Title: Pilot and Feasibility Study of a MAWDS (Medications, Activity, Weight, Diet and Symptoms) Heart Failure Mobile Platform
Acronym: iMAWDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Savvysherpa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1050557
Record Dates: First submitted 2017-09-13; First posted 2017-09-27 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Failure Patients (Experimental): Patients who are seen at Intermountain Medical Center with heart failure, based on the Intermountain-specific Heart Failure Identification and Risk Stratification, will be screened for this study. The Principal Investigator and/or his delegate will confirm the presence of heart failure, based on established standard of care criteria for diagnosis.
  Interventions: Behavioral: MAWDS data entry on app

INTERVENTIONS:
Behavioral: MAWDS data entry on app — Utilize the smartphone app to enter their MAWDS (Medication, Activity, Weight, Diet, Symptoms) data

SUMMARY:
The purpose of this study is to create a smartphone app that delivers the educational content of the current Intermountain MAWDS* program and allows patients to enter and track their MAWDS data within the app; and to determine if a broad-scale project can be conducted within the limits of currently available technology. Information from this study will be used to design a larger study that is powered to assess the association between data obtained via a MAWDS app and heart failure outcomes.

(*MAWDS- Medications, Activity, Weight, Diet, Symptoms)

DETAILED DESCRIPTION:
The Intermountain Heart Institute will collaborate with Savvysherpa Inc to develop a sensor-based digital platform based on MAWDS. (MAWDS is Intermountain's acronym that stands for Medications, Activity, Weight, Diet, Symptoms; used across Intermountain Healthcare to represent the most important concepts and skills to teach heart failure patients) This will be used to deliver simple, home-based interventions via an app on the subject's iPhone. The app will be programmed to send notifications to the subject to enter their MAWDS data and perform a 6-minute walk test at specific time points during the study. Written informed consent will be obtained from each subject prior to participation. A study team member will register eligible subjects as well as assist them with the iPhone and HealthKit set-up and train them on the app usage. Protocol-required information will be obtained from subject's medical records (collected as part of their usual medical care). Subjects will be asked to enter data into the MAWDS iPhone app at specified intervals for a period of 3 months. The data, with the date and time it was entered, will be posted to a study-specific database. Periodically, the MAWDS app will query activity data from HealthKit and post that to the same database. Scheduled notifications will appear in the iPhone's Notification Center, reminding the subject to use the app. To assess subject engagement, the app will collect and store standard usage statistics provided by the iOS (e.g., number of times and duration the app is used per day, number of data entries, etc). The subjects' electronic medical records will be reviewed for a period of 3 months following enrollment, focused on healthcare utilization (e.g., hospital readmissions, mortality, changes in Intermountain HF (heart failure) Risk Score, etc). All information will be made part of the study-specific database. Follow-up phone calls will be done, as needed, within the first 2 weeks after enrollment to remind subjects to activate the app, ensure that the subjects are using the app appropriately, and address any issues noted on monitoring the data collected via the app. Subjects will have no other research-related clinic visits or in-person follow-up evaluations, other than the visit for obtaining informed consent, registration and setting up of the app, and follow-up telephone calls as needed. Upon completion of the study, the app on the subject's iPhone will be disabled and Savvysherpa will disconnect the "backend" data capture. Data will no longer be collected from the subject and his/her medical records will no longer be accessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age
2. Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures
3. Documentation of heart failure of any etiology, using standard of care criteria for diagnosis, and based on clinical assessment of the Principal Investigator and/or his delegate
4. Possess (and are comfortable using) an iPhone of appropriate age (model 5S or newer, since these models have a motion coprocessor that can run iOS 8 or later, as needed to run the app)
5. Willing and able to comply with the instructions for entering their MAWDS data into the app installed in their iPhones

Exclusion Criteria:

1. Significant and/or severe co-morbidities, as assessed by the Principal Investigator and/or his delegate
2. Currently in hospice care or planned discharge to hospice care at home or to a hospice care facility
3. Inability to read and/or understand English (Non-English speaking and reading participants will be excluded since the program requires a variety of communications, not all of which have been validated in a language other than English).
4. Other conditions that in the opinion of the Principal Investigator and/or Sub-Investigator may increase risk to the subject and/or compromise the quality of the clinical trial
5. The Study Clinician(s) determine(s) that the subject is not eligible for participation in this research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
The number of patients utilizing the app. | 3 months
  Data will be collected that shows the number of patients engaging with the app.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk U Knowlton, MD, Principal Investigator — Intermountain Heart Institute
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No